CLINICAL TRIAL: NCT06531096
Title: Optimising Inhaler Technique and Asthma Self-management in Children and Young People
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Dara O'Donoghue, Clinical Senior Lecturer, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 293828
Record Dates: First submitted 2023-12-04; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Asthma in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group- v-DOT (Experimental): The intervention group will have the v-DOT (video directly observed therapy) App downloaded to their Phone or Tablet and will be instructed on how to take and upload audio-videos of themselves or their child taking their inhaler and/or nasal spray.
  The audio videos will be time/date stamped and forwarded to the secure repository. Depending on the prescribed frequency of the preventer asthma and allergic rhinitis inhalers or sprays these audio videos will be uploaded once or twice-daily. These videos will be reviewed every morning by the lead researcher (trained in inhaler and nasal spray technique assessment and training) who will provide feedback via email or an instant messenger service. Videos will be evaluated using an inhaler/ nasal spray checklist.
  The use of v-DOT to upload audio videos with feedback will continue until the patient has uploaded 3 consecutive days of correct technique (up to a maximum of 21 days).
  Interventions: Behavioral: v-DOT
- Control group- standard care (No Intervention): All enrolled patients will have an educational session with an asthma nurse using teach back methodology to teach inhaler and/or nasal spray technique and personalised asthma action plan (PAAP). During this session education is given on what asthma is, identifying and avoiding triggers, asthma treatments, and side effects of treatment.
  The control participants will have further assessment and educational sessions using teach back methodology to ensure correct inhaler technique is mastered and understanding of how to action the three zones of the PAAP until they have achieved 'mastery' of the technique and understanding of their PAAP.

INTERVENTIONS:
Behavioral: v-DOT — Video directly observed therapy
  Arms: Intervention group- v-DOT

SUMMARY:
The aim of this randomised pilot study is to explore ways to optimise a care pathway that results in children and young people with asthma being better trained in the basics of asthma care and better able to apply self-management at the earliest possible stage.

This will involve comparing a novel augmented teaching method (Video directly observed therapy (v-DOT)) with standard training in achieving and sustaining mastery of inhaler and nasal spray technique and the understanding of a personalised asthma action plan (PAAP).

DETAILED DESCRIPTION:
The aim of this randomised pilot study is to explore ways to optimise a care pathway that results in children and young people with asthma being better trained in the basics of asthma care and better able to apply self-management at the earliest possible stage.

This will involve comparing a novel augmented teaching method (Video directly observed therapy (v-DOT)) with standard training in achieving and sustaining mastery of inhaler and nasal spray technique and the understanding of a personalised asthma action plan (PAAP).

Children with acute wheezing referred to the Safe Asthma Discharge Care Pathway (SADCP) service will be approached for participation. Participants will then be randomised 1:1 to either remain in the SADCP (control) or to receive the v-DOT enhancement (intervention).

All enrolled patients will have an educational session with an asthma nurse using teach back methodology to teach inhaler and/or nasal spray technique and personalised asthma action plan (PAAP). During this session education is given on what asthma is, identifying and avoiding triggers, asthma treatments, and side effects of treatment.

The control participants will have a further assessment and educational sessions using teach back methodology to ensure correct inhaler technique is mastered and understanding of how to action the three zones of the PAAP until they have achieved 'mastery' of the technique and understanding of PAAP.

The intervention group will immediately have the v-DOT App downloaded to their phone or tablet and will be instructed on how to take and upload audio-videos of themselves or their child taking their inhaler and/or nasal spray. The use of v-DOT to upload audio videos with feedback will continue until the patient has uploaded 3 consecutive days of correct technique (up to a maximum of 21 days). Reminders will be sent via email if the patient fails to upload any videos for 24 hours to serve as a prompt for uploading the daily videos.

It is not possible to blind either the participants or the assessors due to the nature of the intervention itself. As this is a pilot study, no sample size has been calculated. A convenience sample will be enrolled over the course of 6-9 months.

Mastery of inhaler technique will be defined as absence of healthcare professional detected errors. Inhaler technique and nasal spray technique will be scored on locally agreed checklists, informed by a scoping review on how inhaler technique is assessed in children and young people and reviewed by the local Asthma multidisciplinary team to agree critical steps. These checklists have been adapted to include "critical errors" in the steps. In addition, a global assessment will be made: correct, partially correct and poor technique. Scoring of inhaler technique will be performed independently by two members of the research team to account for inter-observer variability.

All participants (control and intervention) will be followed up at 1 month, 3 months and 6 months after achieving mastery of technique.

Teaching of the unique personalised asthma action plan (PAAP) is an integral part of the teach back process at the safe asthma discharge care pathway service. The investigators will assess new patient's understanding of their PAAP as they enter the SADCP (prior to education) and compare this to their understanding at follow up. The investigators will compare long term PAAP understanding of the control group (who will have received additional teach back sessions) to the intervention group (who will have received only 1 teach back session). The investigators will also compare patient's understanding of their PAAP with clinical outcomes.

In order to determine if v-DOT has promise of being cost effective in comparison to standard care, a within-study cost-effectiveness analysis will be conducted from the provider perspective (health services).

To explore potential reasons for poor inhaler technique, incorrect implementation of personalised asthma action plans and potential barriers encountered and to evaluate the experiences of the participants to determine if they feel that this method of teaching and monitoring technique is acceptable, participants will be invited to participate in semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* 1-15 years of age (up to 16th birthday)
* Established asthmatic children (prescribed an inhaled corticosteroid preventer), who have been admitted or referred for paediatric ward review or attended A&E with their 2nd acute wheeze episode within a 6-month period.
* Established asthmatic children (prescribed an inhaled corticosteroid preventer), with inadequate control whom medical staff feel would benefit from further education.
* 3rd viral induced wheezing episode within 6 months, in those already prescribed an inhaled corticosteroid preventer (but not formally 'asthma').
* English and non-English speaking children and young people will be eligible as we have access to translation services that are already utilised at our asthma clinics.

Exclusion Criteria:

* Children who have previously received intervention through the safe asthma discharge care pathway service.
* < 1 year of age.
* Children and young people with cough but no wheeze.
* Those children who are referred to paediatric asthma clinic or nurse led asthma clinic, where they have received teach back training on inhaler technique/nasal spray technique and PAAP training.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Mastery of technique | Once mastery of technique established which is defined as 3 consecutive days of correct technique.
  Number of days of video directly observed therapy (v-DOT) required to achieve 'mastery' following one initial educational session using teach back methodology for asthma inhaler +/- nasal spray (for those with concomitant allergic rhinitis).
Technique score | Baseline and 1, 3 and 6 months after achieving technique mastery
  Inhaler with or without nasal spray technique at baseline and 1,3 and 6 months after achieving technique mastery. Technique will be scored as a proportion of the correct steps taken (using locally agreed inhaler and nasal spray checklists). Scores range from 0 to 5, with 5 being the maximum and a higher score having a better outcome. This will then be converted to a percentage. Mastery of inhaler technique will be defined as absence of healthcare professional detected errors. The proportion of correct steps taken will be described for each group using descriptive statistical measures. In addition, a global assessment will be made: correct, partially correct and poor technique.
Personalised asthma action plan (PAAP) understanding. | Baseline and 1, 3 and 6 months after achieving technique mastery
  Understanding of their personalised asthma action plan will be measured at baseline and 1,3 and 6 months after achieving technique mastery. This will be assessed by asking questions using a pre-defined checklist to clarify if they know which medications they should take every day and what they should do if they become unwell with regards to their treatment regime.
  Maximum value = 5. Minimum value = 0. A score of 5 means complete understanding of the personalised asthma action plan. A higher score means a better outcome.
Recruitment rates | Through study recruitment, an average of 1 year.
  Recruitment rates and a description of barriers to and how to facilitate.
Retention rates | At study completion for all participants, up to 2 years.
  Patients who complete full follow up and those who withdraw or fail to complete the full study.
Qualitative interviews to identify barriers to using video directly observed therapy (v-DOT) | 3-6 months after achieving mastery of technique.
  Barriers to using video directly observed therapy (v-DOT) for example participation rates, technical considerations, ability to correct inhaler error using v-DOT and use of resources.

SECONDARY OUTCOMES:
Health service resource use and incremental cost-effectiveness. | Through study completion, up to 1 year.
  In order to determine if v-DOT has promise of being cost effective in comparison to standard care, a within-study cost-effectiveness analysis will be conducted from the provider perspective (health services).
Spirometry | At baseline following recruitment to the study and 6 months after achieving mastery of technique.
  Each child who is old enough to perform spirometry in clinic will have their FEV1 and FVC measured using standardised spirometry equipment. The forced expiratory volume in 1 second (FEV1) is the volume of air exhaled in the first second during forced exhalation after maximal inspiration. Forced vital capacity (FVC), the maximum amount of air that can be exhaled when blowing out as fast as possible. Expressed in litres. This will then be converted to a percentage predicted when compared to others of the same sex, height and weight and expressed as a percentage. A higher percentage meaning better outcomes.
Fractional exhaled nitric oxide (FeNO) | At baseline following recruitment to the study and 6 months after achieving mastery of technique.
  Each child who is old enough to perform spirometry in clinic will have their Fractional exhaled nitric oxide (FeNO) measured using standardised equipment. Result expressed as parts per billion. Minimum value of 0. No maximum value cut off defined. A higher value means worse outcomes.
Number of prescribed oral corticosteroids | At baseline following recruitment to the study and 6 months after achieving mastery of technique.
  Number of prescribed oral corticosteroids in previous 12 months prior to recruitment and since achieving mastery of technique.
Number of emergency department and out of hours attendances | At baseline following recruitment to the study and 6 months after achieving mastery of technique.
  Number of emergency department and out of hours attendances with acute wheeze in previous 12 months prior to recruitment and since achieving mastery of technique.
Number of admissions with acute wheeze | At baseline following recruitment to the study and 6 months after achieving mastery of technique.
  Number of admissions with acute wheeze in previous 12 months prior to recruitment and the 6 months since achieving mastery of technique. Including length of stay in hospital.
Adherence to inhaled corticosteroid medication. | At baseline following recruitment to the study and 6 months after achieving mastery of technique.
  Adherence to inhaled corticosteroid medication (as determined by General Practitioner prescription pick-ups) and analysed using the medication refill adherence approach. Medication refill adherence is the total days supply divided by the total number of days of study participation and multiplied by 100 to provide a percentage adherence value. Minimum value is 0% and maximum is 100%. A value of 100% having the best outcome.
Children's asthma control test (c-ACT) score. | At baseline following recruitment to the study and 6 months after achieving mastery of technique.
  A validated questionnaire which is scored from 0 to 27. A higher score has a better outcome. A score of 19 or lower means the child's asthma has not been well controlled.
Mini- paediatric quality of life questionnaire score. | At baseline following recruitment to the study and 6 months after achieving mastery of technique.
  A validated quality of life questionnaire. Scored from 13 (minimum score) to 91 (maximum score). A higher scores means a better outcome/ less impact on their quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dara O'Donoghue, MD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Belfast Health and Social care trust, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No